CLINICAL TRIAL: NCT07066566
Title: The Effect of Asymmetrical vs. Symmetrical High Flow Nasal Cannula on the Work of Breathing: A Randomised Cross-over Study
Brief Title: The Effect of Asymmetrical vs. Symmetrical High Flow Nasal Cannula on the Work of Breathing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Ioannis Pantazopoulos, Associate Professor of Respiratory & Emergency Medicine Faculty of Medicine, University of Thessaly, Greece, Larissa University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16171
Record Dates: First submitted 2025-06-24; First posted 2025-07-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Disease (Clinically Stable Individuals - Patients Recovered From Respiratory Disease)
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery patients from respiratory disease - Asymmetric or conventional nasal high flow cannula (Experimental): Patients recovered from acute respiratory disease will be randomized to NHF oxygen therapy with asymmetrical cannula or conventional cannula
  Interventions: Device: Asymmetric nasal cannula - DUET; Device: Conventional nasal high flow cannula
- Recovery patients from respiratory disease - Conventional or asymmetric nasal high flow cannula (Active Comparator): Patients recovered from acute respiratory disease will be randomized to NHF oxygen therapy with conventional cannula or asymmetrical cannula
  Interventions: Device: Asymmetric nasal cannula - DUET; Device: Conventional nasal high flow cannula

INTERVENTIONS:
Device: Asymmetric nasal cannula - DUET — DUET asymmetric nasal high flow interface that fits best to patients' nostrils (size: one nostril of the patient should be fully occluded) Patients will be crossed - over between the 2 interventions
Device: Conventional nasal high flow cannula — Well - established conventional nasal high flow cannula (size: medium) Patients will be cross - over between the 2 interventions

SUMMARY:
The goal of this study randomized single-center crossover study is to evaluate the impact of asymmetrical versus symmetrical nasal high flow (NHF) therapy on work of breathing (WOB). The main question it aims to answer are:

1. Does the asymmetrical NHF interface improve the work of breathing compared to the symmetrical NHF interface? Researchers will compare the symmetrical NHF interface to the symmetrical NHF interface to see if the the asymmetrical interface has a greater impact on the work of breathing.

Participants will :

1. receive NHF via both interfaces (FiO₂ 0.21, 50 L/min) for 15 minutes, in random order, with esophageal pressure monitoring and bioelectrical impedance analysis performed.
2. baseline characteristics will me monitored throughout the interventions
3. Esophageal pressure and minute ventilation will be monitored.

DETAILED DESCRIPTION:
Each participant will undergo all phases of the study while seated comfortably, breathing room air. Vital signs, including blood pressure, heart rate, and peripheral oxygen saturation (%SpO₂), will be continuously monitored and recorded throughout.

Respiratory mechanics will be assessed using esophageal pressure (Pes) monitoring. A thin latex balloon catheter (10 cm long, 3-5 cm circumference; Cooper surgical, USA), filled with 0.5 mL of air, will be placed in the mid-esophagus (~45 cm from the nares) and will be connected to a pressure transducer (RSS-100HR, Hans Rudolph Inc., USA). Correct positioning will be confirmed by observing equal fluctuations in Pes and airway pressure (Paw) during occluded breaths. Balloon integrity will be verified before, after, and as needed during the procedure.

Participants will be instructed to breathe quietly on room air (FiO₂ 0.21) to allow for baseline assessment. Volume will be recorded using a heated pneumotachometer (Series 3813; Hans Rudolph Inc., USA) and the Research Pneumotach System (RSS100-HR), sampling at 50 Hz, a sampling rate exceeding the Nyquist criterion for respiratory signals. A bioelectrical impedance technology device (ExSpiron, Respiratory Motion Inc., Waltham, MA) will then be attached around the chest to assess lung volume changes.

Participants will then be randomized in a 1:1 ratio to one of two intervention sequences using a computer-generated randomization schedule.

* Sequence 1: Symmetrical NHF Interface - 3-minute washout period - Asymmetrical NHF Interface
* Sequence 2: Asymmetrical NHF Interface - 3-minute washout period - Symmetrical NHF Interface In the seated position, participants will both 15-minute phases, separated by a 3-minute washout period to prevent residual effects. During the "Symmetrical Interface" phase, participants will breathe using the conventional symmetrical NHF cannula, and during the asymmetrical phase, the asymmetrical interface (DUET, Fisher and Paykel Healthcare, Auckland, New Zealand) will be used. High-flow oxygen will be delivered using a commercial system (AIRVO 3; Fisher and Paykel Healthcare, Auckland, New Zealand) set at a flow of 50 L/min, temperature of 37°C, and FiO₂ of 0.21.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years old
2. absence of symptoms and signs of respiratory failure (SpO2>95% at FiΟ2 0.21)

Exclusion Criteria:

1. pregnancy
2. SpO2<94% at FiΟ2 0.21
3. neuromuscular disease
4. contraindications to esophageal pressure monitoring (e.g., uncontrolled coagulopathy, esophageal disease, nasal trauma, allergy to local lidocaine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in the pressure time product after the use of symmetrical high flow nasal interface for 15 minutes. | Baseline and 15 minutes
  This outcome measures the change in the Pressure-Time Product (PTP) before and after the application of a symmetrical high-flow nasal interface (HFNI) in patients requiring noninvasive respiratory support. The PTP is a physiological index that reflects the work of breathing and respiratory muscle effort. It is calculated using airway pressure and inspiratory time data over a defined period. The primary goal is to assess whether the symmetrical HFNI leads to a measurable reduction in the PTP, indicating improved respiratory mechanics and decreased patient effort.
Change in the pressure time product after the use of asymmetrical nasal high flow interface for 15 minutes. | Baseline and 15 minutes
  This outcome measures the change in the Pressure-Time Product (PTP) before and after the application of a symmetrical high-flow nasal interface (HFNI) in patients requiring noninvasive respiratory support. The PTP is a physiological index that reflects the work of breathing and respiratory muscle effort. It is calculated using airway pressure and inspiratory time data over a defined period. The primary goal is to assess whether the asymmetrical HFNI leads to a measurable reduction in the PTP, indicating improved respiratory mechanics and decreased patient effort.

CONTACTS AND LOCATIONS:
Overall Officials: Demosthenes Makris, Study Chair — Professor of Intensive Care Unit, University Hospital of Larissa
Locations (1):
- University Hospital of Larissa, Department of Pulmonary Medicine, Larissa, Greece

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT07066566/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT07066566/ICF_001.pdf